CLINICAL TRIAL: NCT06444659
Title: Effects of Adaptive Physical Activity on Health-related Fitness of Students With Intellectual Disabilities
Brief Title: Effects of Adaptive Physical Activity on Health-related Fitness of Students With Intellectual Disabilitiesdisability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Peiying Huang, Principal Investigator, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HunanNU
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intellectual Disability
Keywords: intellectual disability; health-related Fitness; Fundamental movement skills
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive physical activities (Experimental): 1. Intervention time: 6 months
  2. Exercise frequency: 3 times/week
  3. Exercise type: aerobic exercise
  4. Exercise intensity: 40-80% HRmax
  5. Collaborating with families to create a parent-supported exercise environment
  Interventions: Behavioral: Adaptive Physical Activity Classes
- Traditional physical education (No Intervention): Continue to carry out the original regular physical education activities during the same period of time, and maintain the original daily habits.

INTERVENTIONS:
Behavioral: Adaptive Physical Activity Classes — The intervention group received a 6 months adaptive physical activity intervention; the control group, on the other hand, continued their original regular physical activity programme for the same period of time and maintained their original lifestyle habits.
  Arms: Adaptive physical activities

SUMMARY:
The object of this study is the theory and practice of adaptive physical activity for people with intellectual disability. It focuses on the concepts, paths, and applications of adaptive physical activities for young people with intellectual disability, and systematically studies and discusses the concepts, paths, and application strategies of adaptive physical activities for young people with intellectual disability, so as to provide solutions and support for the scientific exercise of this special population group. The study will focus on the following four aspects: (1) theoretical research on the interventions of young people with intellectual disability (2) analysis of the sports and health needs of young people with intellectual disability (3) empirical research on adaptive physical activities for young people with intellectual disability (4) exploration of strategies for the use of adaptive physical activities.

Based on theoretical and practical research, to understand the current situation of sports participation and influencing factors of Effects of adaptive physical activity on health-related Fitness and Fundamental Movement Skills in students with intellectual disability , to provide a reliable basis for the formulation of adaptive sports activity programmes suitable for the rehabilitation concepts of the Effects of adaptive physical activity on health-related Fitness and Fundamental Movement Skills in students with intellectual disability; to increase the interest of Effects of adaptive physical activity on health-related Fitness and Fundamental Movement Skills in students with intellectual disability in sports activities, so as to enable them to master the basic sports skills, have the physical abilities required for completing the basic social activities, and be able to participate in sports activities on a regular basis in their future lives; and to promote their physical health and happy lives, with a view to facilitating their integration into regular education and, ultimately, social integration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Intellectual disability
* Agree and promise to participate in the exercise intervention throughout the study programme
* No other physical activity other than participation in school sports

Exclusion Criteria:

* Have other medical conditions that limit physical activity (e.g. asthma, heart disease, etc.)
* Suffers from complex neurological disorders
* unable to play sports due to abnormal physical development

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Muscular strength and endurance within Health-Related Physical Fitness are assessed using the handgrip strength test | up to 6 months
Body mass index (BMI) was computed based on measurements of weight and height | up to 6 months
Body fat percentage | up to 6 months
Flexibility was assessed using the Sit-and-Reach test | up to 6 months
Cardiopulmonary fitness was assessed via the 20 m PACER run | up to 6 months
FMS assessment: The Test of Gross Motor Development-2 (TGMD-2) for assessing participants' FMS development | up to 6 months

SECONDARY OUTCOMES:
Objective measurement of participants' sleep quality using the Actigraph GT3X+ | up to 6 months
Physical Activity Leves: ActiGraph GT3X+ (ActiGraph LLC, Pensacola, FL) triaxial accelerometers | up to 6 months
Quality of life : We assessed quality of life (QoL) using the World Health Organization Quality of Life (WHOQOL) scale. | up to 6 months
  Participants responded to 12 items, with each item providing five response options. The total score ranges from 12 to 60, with higher scores indicating better quality of life.
The Physical Activity Enjoyment Scale (PACES): It is used to assess enjoyment of physical activity. | up to 6 months
  The questionnaire consists of 16 questions rated on a 5-point scale. The scale consists of 9 positively worded items and 7 negatively worded items. Scores for the 7 negatively worded items are reverse-coded and then combined with the scores for the positively worded items. Higher total scores indicate greater levels of enjoyment.
Childhood Autism Rating Scale (CARS): It is used to assess the severity of autism symptoms. | up to 6 months
  The CARS consists of 15 items, each addressing different aspects of autism. Each item is rated on a scale from 1 to 4, where 1 indicates "behavior comparable to age expectations," 2 denotes "slightly atypical," 3 reflects "moderately atypical," and 4 signifies "severely atypical." The total score ranges from 15 to 60, with higher scores indicating more severe autism symptoms. Scores between 30 and 37 indicate mild to moderate autism, while scores above 37 represent severe autism.
Sleep Disturbance Scale for Children (SDSC): It is used to evaluate the severity of sleep disturbances. | up to 6 months
  It includes 26 items rated on a 5-point Likert scale from "never" to "always," with scores ranging from 1 to 5. A total score above 39, based on Bruni et al.'s study, indicates sleep disturbances, with a sensitivity of 0.89 and specificity of 0.74.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Physical Education, Hunan Normal University, Changsha, China

REFERENCES:
- [Derived] Shen X, Huang P, Liu Q, Guo Y, Zheng L. Telehealth based parental support over 6 months improves physical activity and sleep quality in children with autism: a randomized controlled trial. Front Pediatr. 2024 Oct 25;12:1496827. doi: 10.3389/fped.2024.1496827. eCollection 2024. PMID 39525834